CLINICAL TRIAL: NCT00032448
Title: CSP #456 - Tension Free Inguinal Hernia Repair: Comparison of Open and Laparoscopic Surgical Techniques
Brief Title: Does Tension-Free Herniorrhaphy or Laparoscopic Herniorrhaphy Achieve Equal or Better Recurrence Rates and Lower Costs While Achieving Equivalent Outcomes for Hernia Patients?
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: American College of Surgeons (Other)
Responsible Party: Neumayer, Leigh - Study Chair, Department of Veterans Affairs
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 456
Record Dates: First submitted 2002-03-20; First posted 2002-03-22 (Estimated); Last update posted 2011-04-14 (Estimated); Status verified 2011-04

CONDITIONS: Hernia
Keywords: Hernia; laparoscopic herniorrhaphy; tension-free herniorrhaphy
MeSH Terms: conditions — Hernia | interventions — Prostheses and Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): Open and laparoscopic herniorrhaphy
  Interventions: Procedure: Standardized tension-free herniorrhaphy with prosthesis

INTERVENTIONS:
Procedure: Standardized tension-free herniorrhaphy with prosthesis — Compare the effect of two typs of operative treatment of inguinal hernia.

SUMMARY:
Inguinal hernia is one of the most common worldwide afflictions of men. The presence of an inguinal hernia is indication for its repair. Approximately 700,000 hernia repairs are performed in the U.S. each year, and this procedure accounts for 10% of all general surgery procedures in the Veterans Health Administration (VHA) (10,000 inguinal herniorrhaphies performed per year). There are many different techniques currently in use for repairing inguinal hernias and with the advent of laparoscopy, yet another technique is being advocated. Laparoscopic repair has been reported in some studies to be superior to open repair because of less pain and earlier return to work. However, laparoscopic repair requires a general or regional anesthetic and expensive equipment and supplies to perform. There is also evidence that open tension-free mesh repair may have results similar to laparoscopic repair for these patient centered outcome measures. The general acceptance of this procedure, especially in the VHA, has not been uniform. Furthermore, no randomized trial of sufficient size and power to be conclusive has been done to set forth the operative "gold standard" for hernia repair.

DETAILED DESCRIPTION:
Primary Hypothesis: Open tension-free herniorrhaphy when compared with laparoscopic herniorrhaphy will achieve equal or better recurrence rates and lower costs while achieving equivalent outcomes for patient-centered measures.

Secondary Hypotheses:

Intervention: Patients randomized to open repair will undergo a standardized tension-free herniorrhaphy with prosthesis (method of Lichtenstein). Patients randomized to laparoscopic herniorrhaphy will undergo a standardized preperitoneal repair with prosthesis, using either a transperitoneal or extraperitoneal approach. During the implementation period of the trial, a preliminary laboratory session will be conducted with all site PIs to standardize herniorrhaphy techniques, reach consensus on all aspects of perioperative patient management (including postoperative patient instructions, follow-up schedules, definitions of recurrence and complications), and to ensure that the site PI is thoroughly familiar with the protocol.

Each site will be visited by one of two expert surgeons (the Study Chair or a Co-PI surgeon) to observe the operative procedures and ensure that participating surgeons adhere to the protocol in all respects. The first visit will take place in the first 6 months of the study and then as needed thereafter, based on routine examination of operative records randomly selected from each site (5 open and 5 laparoscopic herniorrhaphies, and, if appropriate, viewing of videotapes of the laparoscopic procedures).

Primary Outcomes: Hernia recurrence rate.

Study Abstract:

Background: Inguinal hernia is one of the most common worldwide afflictions of men. The presence of an inguinal hernia is indication for its repair. Approximately 700,000 hernia repairs are performed in the U.S. each year, and this procedure accounts for 10% of all general surgery procedures in the Veterans Health Administration (VHA) (10,000 inguinal herniorrhaphies performed per year). There are many different techniques currently in use for repairing inguinal hernias and with the advent of laparoscopy, yet another technique is being advocated. Laparoscopic repair has been reported in some studies to be superior to open repair because of less pain and earlier return to work. However, laparoscopic repair requires a general or regional anesthetic and expensive equipment and supplies to perform. There is also evidence that open tension-free mesh repair may have results similar to laparoscopic repair for these patient centered outcome measures. The general acceptance of this procedure, especially in the VHA, has not been uniform. Furthermore, no randomized trial of sufficient size and power to be conclusive has been done to set forth the operative gold standard for hernia repair.

Objectives: To determine whether open tension-free herniorrhaphy when compared with laparoscopic herniorrhaphy can achieve equal or better recurrence rates and lower costs while achieving equivalent outcomes for patient-centered measures.

Methods: This multi-center VA cooperative study is enrolling 2200 men with inguinal hernia and randomizing them to one of two operative techniques: open tension-free (Lichtenstein) repair, or laparoscopic preperitoneal repair. The primary outcome measure is recurrence at two years. Secondary outcome measures are complications, pain, time to return to normal activities, health-related quality of life, patient satisfaction, caregiver burden, and cost. The role of comorbidity in the outcome will also be determined. The sample size will permit at least 80% power to detect a difference of 3% in 2-year recurrence rates between the two surgical procedures. Fourteen VAMCs are randomizing the 2200 patients over a 3-year accrual period. The study will also have a 2-year follow-up period. All patients will be followed to the end of the study so that follow-up will range from 2-5 years (average 3.5 years).

On November 29, 2001, the Hines Cooperative Studies Human Rights Committee and the Data and Safety Monitoring Board met to review the data from CSP #456. Both committees determined that there were sufficient data to complete the trial without enrolling any additional patients and recommended that enrollment be stopped. There were no safety concerns. Approximately 2,165 patients of a targeted 2,200 had been enrolled at this point. All sites were notified of this within 24 hours of the action.

Main Manuscript:

ELIGIBILITY:
Inclusion Criteria:

Men with inguinal hernia.

Exclusion Criteria:

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2200 (Estimated)
Dates: Start 1998-10; Primary Completion 2003-12 (Actual); Study Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
To assess recurrence rates, operative complications, pain, convalescent time, health-related quality of life, patient satisfaction, and health care utilization and costs. | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Leigh A. Neumayer, Study Chair — VA Salt Lake City Health Care System, Salt Lake City
Locations (14):
- United States (14):
  - VA Medical Center, Birmingham, Birmingham, Alabama
  - Central Arkansas VHS Eugene J. Towbin Healthcare Ctr, Little Rock, No. Little Rock, Arkansas
  - VA Medical Center, San Francisco, San Francisco, California
  - VA Greater Los Angeles Healthcare System, West LA, West Los Angeles, California
  - James A. Haley Veterans Hospital, Tampa, Tampa, Florida
  - VA Maryland Health Care System, Baltimore, Baltimore, Maryland
  - VA Medical Center, Jamaica Plain Campus, Boston, Massachusetts
  - John D. Dingell VA Medical Center, Detroit, Detroit, Michigan
  - VA Medical Center, Durham, Durham, North Carolina
  - WJB Dorn Veterans Hospital, Columbia, Columbia, South Carolina
  - VA Medical Center, Memphis, Memphis, Tennessee
  - VA North Texas Health Care System, Dallas, Dallas, Texas
  - Michael E. DeBakey VA Medical Center (152), Houston, Texas
  - VA Salt Lake City Health Care System, Salt Lake City, Salt Lake City, Utah

REFERENCES:
- [Result] Neumayer L, Giobbie-Hurder A, Jonasson O, Fitzgibbons R Jr, Dunlop D, Gibbs J, Reda D, Henderson W; Veterans Affairs Cooperative Studies Program 456 Investigators. Open mesh versus laparoscopic mesh repair of inguinal hernia. N Engl J Med. 2004 Apr 29;350(18):1819-27. doi: 10.1056/NEJMoa040093. Epub 2004 Apr 25. PMID 15107485